CLINICAL TRIAL: NCT03748446
Title: Xenon Inhalation Therapy for Major Depressive Disorder and Bipolar Disorder
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Andrew A. Nierenberg, MD, Principle Investigator, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018P002500
Record Dates: First submitted 2018-11-19; First posted 2018-11-20 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Major Depressive Disorder; Bipolar Depression
MeSH Terms: conditions — Depressive Disorder, Major; Bipolar Disorder | interventions — Xenon; Nitrogen

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind crossover model that will compare the effects of xenon-oxygen (35:65 ratio by volume) added to treatment as usual (X-TAU group) to the effects of nitrogen-oxygen (35:65 ratio by volume) added to treatment as usual (N-TAU group). A total of 20 severely depressed patients, 10 with major depressive disorder (MDD) and 10 with Bipolar Depression (BP), will be exposed in random order to N-TAU and X-TAU in a double-blind protocol.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The identity of the inhalant will be blinded to all except the anesthesiologist, who will not participate in any assessment of the depressive symptoms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- X-TAU (xenon) (Active Comparator): Xenon is a potent antiglutaminergic agent that has been used as an anesthetic with minimal side effects, has neuroprotective effects consistent with antidepressants and has the potential to be a novel antidepressant drug.
  - xenon-oxygen (35:65 ratio by volume) added to treatment as usual (X-TAU group)
  Interventions: Drug: Xenon
- N-TAU (nitrogen-placebo) (Placebo Comparator): Nitrogen-oxygen (35:65 ratio by volume) added to treatment as usual (N-TAU group)
  Interventions: Drug: Nitrogen gas

INTERVENTIONS:
Drug: Xenon — The investigators have chosen to use as a maximum concentration about half the general anesthetic partial pressure of xenon (35%=70%/2) to achieve a dose that is sub-anesthetic. This concentration of xenon is very close to that at which subjects emerging from xenon anesthesia first respond to verbal commands, commonly referred to as MAC awake.
  Arms: X-TAU (xenon)
Drug: Nitrogen gas — nitrogen-oxygen (35:65 ratio by volume) added to treatment as usual
  Arms: N-TAU (nitrogen-placebo)

SUMMARY:
The investigators will test the hypothesis that inhaled xenon will produce a rapid improvement in depressive symptoms in patients suffering from treatment-resistant depression. Specifically, the investigators will conduct a parallel randomized, double-blind crossover study that will compare the effects of xenon-oxygen (35:65 ratio by volume) added to treatment as usual (X-TAU group) to the effects of nitrogen-oxygen (35:65 ratio by volume) added to treatment as usual (N-TAU group). A total of 20 severely depressed patients, 10 with major depressive disorder (MDD) and 10 with Bipolar Depression (BP), will be exposed in random order to N-TAU and X-TAU in a double-blind protocol.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) occurs in up to 17% of the population, is associated with profound dysfunction and, according to the WHO Global Burden of Disease Study, is estimated to become the second leading cause of disability worldwide by 2020. While antidepressants have proven efficacy, they usually take weeks to work and then only about a third of patients reach remission.

Beyond the traditional monoaminergic approaches, recent advances in understanding the pathophysiology of MDD have focused on the dysregulation of glutamate and associated neuronal glutaminergic associated excitotoxicity. Xenon is a potent antiglutaminergic agent that has been used as an anesthetic with minimal side effects, has neuroprotective effects consistent with antidepressants, and has the potential to be a novel antidepressant drug.

Although mania or hypomania are the defining characteristics of bipolar disorder, throughout the course of the illness depressive symptoms are more common than manic symptoms. People with bipolar disorder spend a substantial proportion of time with syndromal or subsyndromal depressive symptoms. The risk of suicide is greatly elevated during depressive episodes. Approximately 17% of people with bipolar I disorder and 24% with bipolar II disorder attempt suicide during the course of their illness. Annually around 0.4% of people with bipolar disorder will die by suicide, which is vastly greater than the international population average of 0.017%.

Pharmacological treatments are commonly used during episodes of mania and bipolar depression. Over time these episodes, particularly depression, tend to become more frequent and as repeated episodes are associated with increased functional impairment, effective treatment is a priority. The treatment of bipolar depression is quite challenging. Treatments used during acute episodes include antidepressants, some antipsychotic drugs such as quetiapine, the anticonvulsant drug lamotrigine and lithium. Response to these agents both acutely and during maintenance treatment is often partial. There are concerns about the potential for switching into mania and more frequent cycling mood with antidepressant treatment.

Only a handful of treatments are approved for bipolar depression and have been shown to be superior to placebo (lurasidone, valproate, quetiapine, the combination of fluoxetine and olanzapine, olanzapine alone, and lamotrigine), however atypical antipsychotics carry significant burden of side effects in particular metabolic.

Ketamine has been shown to be efficacious and well tolerated in MDD and BP depression, with low risk of inducing manic switch; other glutamatergic agents like memantine or lamotrigine are used as augmentation in depression and are well tolerated. Therefore, investigators believe Xenon could be well tolerated both in MDD and BP depression and possibly helpful in alleviating the symptoms.

The investigators hypothesize that patients with a primary diagnosis of depression will have a greater decrease in depressive symptoms after one session of xenon inhalation added to treatment as usual (X- TAU) compared to their session with nitrogen-oxygen inhalation added to treatment as usual (N-TAU). The investigators will specifically randomize the 20 patients to receive in random order one session of X- TAU and one session of N-TAU. Blind ratings of depression will be done with the modified Hamilton Depression Rating Scale (HDRS) and Quick Inventory of Depressive Symptomatology-Clinician Version (QIDS-C) at baseline and at predefined time intervals by clinicians experts in mood disorder who will be completely blinded to all the administration procedures.

The methods for depression assessments will be consistent with those used for the early proof-of-concept ketamine studies with assessments at 40, 80, 110, and 230 minutes post-administration and 1, 3, and 7 days post-administration. The primary outcome will be improvement at day 1. Mixed model repeated measures analysis will be used to compare the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Patient who meets DSM-V Criteria for MDD or Bipolar Depression (according to DSM-V), as the primary focus of treatment.
* Able to understand the risks and benefits of participating in this clinical trial and give informed consent, per judgment of the investigator.
* Age greater than or equal to 18 years but less than or equal to 65 years.
* Montgomery Asberg Depression Rating Scale ≥20.
* On an adequate antidepressant regimen (MDD) or on a mood stabilizing regimen (BP) that is stable for at least four weeks prior to enrollment.
* Has reliable adult transportation from and to home.
* Has a treating psychiatrist who is in agreement with the patient's participation in the study, and aware of the safety plan in the protocol.
* No medical contraindications to receiving a xenon- or a nitrogen-oxygen mixture.
* No serious or active pulmonary disease.

Exclusion Criteria:

* MDD or BP disorder with psychosis, schizophrenia, OCD, or a primary anxiety disorder.
* Currently taking a benzodiazepine (including PRN).
* Unwilling or unable to comply with study procedures.
* Active substance abuse in the past 60 days, diagnosis of substance dependence in the past 12 months, currently active smokers of any substance, including prescription marijuana.
* Pregnant women or women of child bearing potential who are not using a medically accepted means of contraception.
* Any unstable medical illness (cardiovascular, hepatic, renal, respiratory, endocrine, neurological, or hematological disease or uncontrolled seizure disorder).
* Any history of brain injury and any active state involving entrapped air/gas within a body cavity with the potential to expand causing organ distension/compression (e.g., bowel obstruction, pneumothorax, or pneumocephalus).
* History of hypersensitivity to xenon; history of multiple adverse drug reactions.
* Have taken any investigational psychotropic drug within the last 6 months.
* Inability to agree to comply with the visit schedule or study procedures.
* Not appropriate for participation in a research trial per judgment of the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-12-05 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Depressive Symptoms | Improvement at day 1
  Hamilton Depression Rating Scale (HDRS):This scale is a 6-item survey which is one of the most frequently used instruments for evaluating depression in adults, the questionnaire allows clinicians to assess the nature and severity of mood disorders in patient populations.
  Score Range: 0-42, higher scores means worse outcomes
Depressive Symptoms | Improvement at day 1
  Quick Inventory of Depressive Symptomatology-Clinician Version (QIDS-C): The Quick Inventory of Depressive Symptomatology (QIDS) is designed to assess the severity of depressive symptoms. The questions to be administered by the clinician assess the severity of the nine diagnostic symptom criteria used in DSM.
  Score Range: 0-48, higher scores means worse outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Nierenberg, MD, Principal Investigator — Massachussetts General Hospital
Locations (1):
- Dauten Family Center for Bipolar Treatment Innovation, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bedi A, McCarroll C, Murray JM, Stevenson MA, Fee JP. The effects of subanaesthetic concentrations of xenon in volunteers. Anaesthesia. 2002 Mar;57(3):233-41. doi: 10.1046/j.0003-2409.2001.02455.x. PMID 11879212
- [Background] Gaynes BN, Warden D, Trivedi MH, Wisniewski SR, Fava M, Rush AJ. What did STAR*D teach us? Results from a large-scale, practical, clinical trial for patients with depression. Psychiatr Serv. 2009 Nov;60(11):1439-45. doi: 10.1176/ps.2009.60.11.1439. PMID 19880458
- [Background] Goto T, Nakata Y, Ishiguro Y, Niimi Y, Suwa K, Morita S. Minimum alveolar concentration-awake of Xenon alone and in combination with isoflurane or sevoflurane. Anesthesiology. 2000 Nov;93(5):1188-93. doi: 10.1097/00000542-200011000-00009. PMID 11046204
- [Background] Kendall T, Morriss R, Mayo-Wilson E, Meyer TD, Jones SH, Oud M, Baker MR. NICE guidance on psychological treatments for bipolar disorder. Lancet Psychiatry. 2016 Apr;3(4):317-20. doi: 10.1016/S2215-0366(16)00082-1. No abstract available. PMID 27063379
- [Background] Kessler RC, Berglund P, Demler O, Jin R, Koretz D, Merikangas KR, Rush AJ, Walters EE, Wang PS; National Comorbidity Survey Replication. The epidemiology of major depressive disorder: results from the National Comorbidity Survey Replication (NCS-R). JAMA. 2003 Jun 18;289(23):3095-105. doi: 10.1001/jama.289.23.3095. PMID 12813115
- [Background] Krystal JH, Karper LP, Seibyl JP, Freeman GK, Delaney R, Bremner JD, Heninger GR, Bowers MB Jr, Charney DS. Subanesthetic effects of the noncompetitive NMDA antagonist, ketamine, in humans. Psychotomimetic, perceptual, cognitive, and neuroendocrine responses. Arch Gen Psychiatry. 1994 Mar;51(3):199-214. doi: 10.1001/archpsyc.1994.03950030035004. PMID 8122957
- [Background] Kupfer DJ, Frank E, Phillips ML. Major depressive disorder: new clinical, neurobiological, and treatment perspectives. Lancet. 2012 Mar 17;379(9820):1045-55. doi: 10.1016/S0140-6736(11)60602-8. Epub 2011 Dec 19. PMID 22189047
- [Background] Ma D, Wilhelm S, Maze M, Franks NP. Neuroprotective and neurotoxic properties of the 'inert' gas, xenon. Br J Anaesth. 2002 Nov;89(5):739-46. PMID 12393773
- [Background] Yonas H, Grundy B, Gur D, Shabason L, Wolfson SK Jr, Cook EE. Side effects of xenon inhalation. J Comput Assist Tomogr. 1981 Aug;5(4):591-2. doi: 10.1097/00004728-198108000-00029. PMID 7264006